CLINICAL TRIAL: NCT06089694
Title: Crome/Cobalt Respiration Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT22030
Record Dates: First submitted 2023-10-09; First posted 2023-10-18 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All Enrolled Subjects: In-clinic Testing Visit: All enrolled subjects will have a Holter recorder, capnography monitor and SpO2 sensor applied and will undergo various breathing/exercise activities. Subjects will go home connected to the Holter recorder for 24 hours for collection of ambulatory data.
  Interventions: Device: Enabling Sensor Research Holter Mode feature

INTERVENTIONS:
Device: Enabling Sensor Research Holter Mode feature — The Sensor Research Holter Mode feature within the Crome and Cobalt ICD and CRT-D devices will be enabled for a short period of time at the In-clinic Testing Visit to allow for desired data collection.

SUMMARY:
The goal of this study is to compare measured respiration rates in various subject scenarios and use conditions between capnography and the Crome and Cobalt ICD and CRT-D MRI SureScan devices (derived using a Holter recorder).

DETAILED DESCRIPTION:
This study will enroll subjects who have already received a Medtronic Crome or Cobalt ICD or CRT-D MRI SureScan device and who meet all of the inclusion criteria and none of the exclusion criteria. Subjects will be asked to complete various breathing/exercise activities while connected to a capnography monitor and a Holter recorder and respiration rates from both devices will be compared for accuracy, with the capnography monitor being the source of truth.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has an active CromeTM or CobaltTM ICD or CRT-D MRI SureScanTM system which has been implanted for at least 30 days and which has not yet reached the Recommended Replacement Time (RRT)
2. Subject is implanted with one of the following models of a true bipolar right ventricular lead manufactured by Medtronic:

   * Model 6946M
   * Model 6947
   * Model 6947M
   * Model 6935
   * Model 6935M
3. Subject is ≥ 18 years of age
4. Subject (or subject's legally authorized representative) is willing and able to provide written informed consent
5. Subject is willing and able to comply with study procedures

Exclusion Criteria:

1. Subject has existing condition that necessitates the use of supplemental oxygen
2. Subject has active acute respiratory infection or respiratory disorder that may affect ability to perform breathing or exercise activities, as assessed by the investigator
3. Any concomitant condition that might endanger the subject through participation in the study or interfere with study procedures, as assessed by the investigator
4. Subject has an active or suspected lead integrity issue, in the opinion of the investigator
5. Subject is enrolled in another study that could confound the results of this study
6. Subject has NYHA Class IV heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study will include adult subjects who are ≥18 years of age, who have an active, implanted Crome or Cobalt ICD or CRT-D system that's been implanted for at least 30 days and which has not yet reached the Recommended Replacement Time (RRT), and who do not have any contraindications that would impact their ability to complete the required breathing and exercise activities, which aligns with the key eligibility criteria for the study. A minimum of 30% of all enrolled subjects will have a documented history of heart failure and a minimum of 20% of all enrolled subjects will be female (as identified at birth).
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Respiration Rates Comparison (Activities Representative of Nightly Average) | During In-clinic Testing Visit, an average of 2 hours
  Difference between the daily respiration rate determined using capnography and the daily respiration rate determined by the Crome and Cobalt ICD and CRT-D devices.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Hartford Hospital, Hartford, Connecticut
  - CentraCare Heart & Vascular Center, Saint Cloud, Minnesota
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas

IPD SHARING:
Plan to Share IPD: No